CLINICAL TRIAL: NCT01041196
Title: Laparoscopic Revision Gastric Bypass Surgery for Perforated Marginal Ulcer: A 10 Year Experience
Brief Title: Perforated Marginal Ulcer After Gastric Bypass
Acronym: PerforatedMU
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Kelvin D Higa, MD; FACS; FASMBS; Professor of Surgery, University of California San Francisco, UCSF Fresno / ALSA Medical Group, Inc. Minimally Invasive Surgery Program
Other Study IDs: CMC IRB No. 2008091; U1111-1113-0006 (Other: World Health Organization, Universal Trial Number)
Record Dates: First submitted 2009-12-26; First posted 2009-12-31 (Estimated); Last update posted 2010-01-01 (Estimated); Status verified 2009-12

CONDITIONS: Ulcer Disease After Gastric Bypass; Marginal Ulcer; Perforated Marginal Ulcer; Acutely Perforated Marginal Ulcer
Keywords: obesity; ulcer disease; marginal ulcer; perforation; abdominal pain; bariatric surgery; weight loss surgery
MeSH Terms: conditions — Peptic Ulcer; Obesity; Abdominal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- perforated ulcer after gastric bypass

SUMMARY:
A common late complication after gastric bypass surgery is marginal ulceration that is defined as ulcers at the margins of the gastrojejunostomy, mostly on the jejunal side. Most marginal ulcers respond to medical therapy and complicated or complex ulcer disease warrants operative intervention; specifically, perforated, penetrated, obstructing, bleeding and intractable marginal ulcers require surgical intervention.

Diverse operative strategies for addressing perforated marginal ulcers after gastric bypass have been described including I) Omental (Graham) patch repair, II) Revision of gastrojejunostomy, III) Irrigation and drainage, IV) any previous procedure with truncal vagotomy, V) Esophagojejunostomy, and VI) Reversal. We formally analyze our experience with the laparoscopic resection and repair of acutely perforated marginal ulcers after Roux-en-Y gastric bypass (RYGB), with or without concomitant resolution of technical risk factors for marginal ulceration.

DETAILED DESCRIPTION:
The epidemic of overweight and obesity in the United States of America along with its comorbidities continues to expand. Bariatric surgery has demonstrated to be the most effective and sustained method to control severe obesity and its comorbidities. For instance, type 2 diabetes mellitus was completely resolved in 76.8%, systemic arterial hypertension was resolved in 61.7%, dyslipidemia improved in 70% and obstructive sleep apnea-hypopnea syndrome was resolved in 85.7%. Furthermore, bariatric surgery significantly increases life expectancy (89%) and decreases overall mortality (30-40%), particularly deaths from diabetes, heart disease, and cancer. Lastly, preliminary evidence about downstream savings associated with bariatric surgery offset the initial costs in 2 to 4 years.

Since 2000, there has been a substantially progressive increase in bariatric surgery. In 2007, the ASMBS reported that 205,000 people had bariatric surgery in the United States from which approximately 80% of these were Gastric Bypass. Moreover, there is a mismatch between eligibility and receipt of bariatric surgery with just less than 1% of the eligible population being treated for morbid obesity through bariatric surgery. Along with the increasing number of elective primary weight loss procedures, up to 20% of post RYGB patients cannot sustain their weight loss beyond 2 to 3 years after the primary bariatric procedure. Thus, revisional surgery for poor weight loss and re-operations for technical or mechanical complications will rise in a parallel manner.

A common late complication after gastric bypass surgery is marginal ulceration that is defined as ulcers at the margins of the gastrojejunostomy, mostly on the jejunal side. Its incidence after RYGB ranges from as low as 0.6 to as high as 16%. After 1,040 laparoscopic RYGB surgeries, the incidence rate, in our hands, is 1.4% and mainly related to NSAID´s use. In observational cohort studies, the presence of specific technical factors - staple-line dehiscence or gastro-gastric fistula, enlarged pouch, foreign material and local ischemia - and environmental factors - tobacco, NSAID´s, alcohol consumption, and H pylori infection among others - have been associated with marginal ulceration however the exact etiopathogenesis has not been completely elucidated.

Similar to peptic ulcer disease, most marginal ulcers respond to medical therapy and complicated or complex ulcer disease warrants operative intervention. Specifically, perforated, penetrated, obstructing, bleeding and intractable marginal ulcers require surgical intervention.

The intestinal mucosa is not typically exposed to gastric acid, which is neutralized by the alkaline biliopancreatic secretions. The jejunal mucosa has no natural barriers; when exposed to gastric acid, it ulcerates easily. Capella & Capella demonstrated that transecting the gastric segments significantly reduce staple-line dehiscence; this is the so-called divided gastric bypass. The incidence for gastro-gastric fistula (GGF) formation after undivided gastric bypass (GBP) was 23%, after a partially divided GBP was 19%, after a completely divided GBP was 2% and after complete transection with interposition of the jejunal limb was 0% (p <0.001).

An unusually large gastric pouch (such as horizontal pouches, retained fundus, long lesser curvature based pouches or enlarged after initially being sized adequately) contain more acid-producing parietal cells. Increased acid production in the pouch carries the risk of developing marginal ulcers. Acid secretion in the small pouch after RYGB is virtually absent.

The anastomotic techniques influence the incidence of marginal ulcers. Capella & Capella reported a consecutive series with significant decrement from 5.1% to 1.5% (p< 0.001) after switching from a stapled to a hand-sewn anastomosis. Likewise, after changing from an inner layer of absorbable suture and an outer layer of nonabsorbable material to a double-layer of absorbable suture the incidence rate improved from 1.6% to 0%.

Local ischemia, in the immediate postoperative period, is probably secondary to technical reasons. Fundamental aspects for decreasing tension and local ischemia at the gastrojejunostomy are dissection of the tissues around the pouch without devascularizing the lesser curvature and complete mobilization of a well-perfused Roux limb.

NSAID´s inhibit prostaglandin synthesis 1) decreasing blood flow to the mucosa (mainly by PG subgroups E and I, which promotes vasodilatation), 2) increased adherence of neutrophils, 3) topical irritant effect, 4) impair of the repair/healing process, and 5) gastric-acid-related effects. In a retrospective cohort study, Wilson et al found NSAID´s consumption to correlate with the marginal ulcer development after RYGB. Numerous studies have identified NSAID´s use as a main risk factor for PUD; however, the precise relevance of NSAID´s as a factor in marginal ulcer development after RYGB is largely unknown.

In epidemiological, clinical and experimental studies, Tobacco has been identified as a major risk factor for peptic ulcer disease (PUD). Smoking carries an overall relative risk of 2.2 for developing PUD. A synergistic relationship for developing PUD exists between H pylori infection and smoking (2.3 vs. 6.1). Biological evidence suggests that smoking compromises the gastric mucosa barrier, decreases gastric emptying and increases gastric secretion. For marginal ulcer after RYGB, there are three cohort studies that showed positive correlation between smoking with developing anastomotic ulcer.

Helicobacter pylori (H pylori) infection carries an overall relative risk of 3.3 (95%CI, 2.6-4.4) for developing PUD. A synergistic relationship exists between H pylori infection and NSAID´s consumption for developing PUD with an overall risk of 3.5 (95%CI, 1.26-9.96) compared to either H pylori or NSAID´s negative individuals. Furthermore, a 61.1 (95%CI, 9.98-373) overall risk exist when compared to H pylori negative individuals not taking NSAID´s. For marginal ulcers after RYGB, three cohort studies have showed that H. pylori infection is not associated with the development of marginal ulcers. In Papasavas et al study, preoperative H. pylori testing with prophylactic eradication did not decrease the incidence of MU or erosive pouch gastritis.

The pathophysiological mechanisms of damage to the gastric mucosa of Ethanol and alcoholic beverages are poorly understood. There are scant retrospective epidemiological studies that determine if a relationship between alcohol consumption and PUD exists. Although alcohol is not associated with an increased risk of PUD, patients with PUD are advised to avoid alcoholic drinks. Basic science studies have showed that instillation of pure ethanol at lower concentrations (4-40% v/v) causes hemorrhagic gastritis in a dose-dependant fashion. Also a synergistic relationship exists between ethanol and NSAID´s, since both cause mucosal injury. On the other hand, there are no studies available about the effect of alcohol on marginal ulcer development after RYGB.

Cocaine use is responsible for approximately 143,000 Emergency Department visits annually; 19% of American, between 18 to 25 years old, have used cocaine: more than 1% of the Americans use cocaine at least once a week; and approximately 50% of all drug-related deaths were secondary to Cocaine. The temporal association between smoking cocaine (crack) and GI tract manifestations include ulceration, perforation, visceral infarction, and retroperitoneal fibrosis. Most ulcer perforations are juxtapyloric or duodenal (D1) however jejunal location has been reported. The physiopathologic hypothesis includes the following mechanisms 1) cocaine blocks the re-uptake of norepinephrine leading to intense vasoconstriction (alpha-adrenergic receptors), mesenteric ischemia, focal tissue ischemia, coagulative necrosis and perforation; and 2) cocaine causes thrombus formation and platelet aggregation mediated by endogenous Thromboxane B2. A few retrospective cohort studies suggest that primary patch repair is the recommended therapeutic option for this type of ulcers. However, Shuster et al reported a high recurrence rate (42%) after omental patch repair compared to a definitive anti-ulcer procedure (0%). Little information exists about the association between crack and gastroduodenal ulcer perforations other than the temporal association reported in small retrospective cohort studies. In a communication, Dr Mason recalls two patients with perforated "stomach ulcers" associated with cocaine use.

The following Critically-Ill patients have a significant increased risk of stress-related mucosal disease (SRMD): 1) mechanical ventilation > 48hrs conveys a 16-fold risk (p < 0.001), 2) coagulopathy has a 4-fold risk (p < 0.001), 3) shock carries a 3.7-fold risk (p= 0.08), 4) drop of intramural pH (from 8 to 6, 5), 5) increase of the number of risk factors (from 0 to 4), 6) recent major surgery, 7) major trauma, 8) severe burns, 9) head trauma, 10) hepatic or renal disease at admission, and 11) sepsis. SRMD encompasses stress-related injury (SRI), which is primarily erosion in the GI tract, and stress ulcer, which is a focal deep mucosal damage. The pathogenesis of SRMD has not being unraveled completely but there is strong evidence that hypoperfusion and reperfusion of the upper GI tract is the major cause. There is no literature available about marginal ulcer after RYGB associated to ICU or critically ill patients.

Diverse operative strategies for addressing perforated marginal ulcers after gastric bypass have been described including I) Omental (Graham) patch repair, II) Revision of gastrojejunostomy, III) Irrigation and drainage, IV) any previous procedure with truncal vagotomy, V) Esophagojejunostomy, and VI) Reversal.

Summarizing, there is scant information about late complications after gastric bypass especially after the widespread adoption of the laparoscopic approach and the modern anatomical construct of Roux-en-Y Gastric Bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic repair of perforated marginal ulcer after RYGB

Exclusion Criteria:

* Perforated marginal ulcers after other bariatric procedures
* Repair by open approach
* Missing records and/or unreachable patients with scant information for analysis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent laparoscopic repair of perforated marginal ulcer after Roux-en-Y gastric bypass (RYGB) for weight loss.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-01; Primary Completion 2009-01 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Morbidity and mortality | at discharge, 1 week, 3 weeks, 8 weeks, 3 months, 6 months, 1 year and annually thereafter for up to 8 years
Recurrence, marginal ulcer. | at 6 months, 1 year and annually thereafter for up to 8 years
Weight loss expressed as Body Mass Index and Percentage of excess weight loss | at 6 months, 1 year and annually thereafter for up to 8 years
Remission or improvement of symptoms | at 6 months, 1 year and annually thereafter for up to 8 years

SECONDARY OUTCOMES:
Remission or improvement of comorbidities | at 6 months, 1 year, and annually thereafter for up to 8 years
Length of operative time which is defined as the time duration of operation measured in minutes from the first skin incision to the final closure of the skin incision | It is measured in minutes from the first skin incision to the final closure of the skin incision at the time of revisional surgery under study. It is a transoperative measure of outcome of the surgery under study
Length of Hospital Stay which is a measured of surgical recovery quantified and reported in days. It is a hospital pre-discharge traditional measure of outcome. | It is measured in days from the admission date to the discharge date for the hospitalization pertaining to revisional surgery under study.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Tercero, MD, Study Director — Research Associate, University of California San Francisco; Kelvin D Higa, MD, Principal Investigator — Professor of Surgery, University of California San Francisco
Locations (1):
- UCSF Fresno Center for Medical Education and Research, Fresno, California, United States

REFERENCES:
- [Background] Higa KD, Boone KB, Ho T, Davies OG. Laparoscopic Roux-en-Y gastric bypass for morbid obesity: technique and preliminary results of our first 400 patients. Arch Surg. 2000 Sep;135(9):1029-33; discussion 1033-4. doi: 10.1001/archsurg.135.9.1029. PMID 10982506
- [Background] Hedley AA, Ogden CL, Johnson CL, Carroll MD, Curtin LR, Flegal KM. Prevalence of overweight and obesity among US children, adolescents, and adults, 1999-2002. JAMA. 2004 Jun 16;291(23):2847-50. doi: 10.1001/jama.291.23.2847. PMID 15199035
- [Background] McTigue KM, Harris R, Hemphill B, Lux L, Sutton S, Bunton AJ, Lohr KN. Screening and interventions for obesity in adults: summary of the evidence for the U.S. Preventive Services Task Force. Ann Intern Med. 2003 Dec 2;139(11):933-49. doi: 10.7326/0003-4819-139-11-200312020-00013. PMID 14644897
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Christou NV, Sampalis JS, Liberman M, Look D, Auger S, McLean AP, MacLean LD. Surgery decreases long-term mortality, morbidity, and health care use in morbidly obese patients. Ann Surg. 2004 Sep;240(3):416-23; discussion 423-4. doi: 10.1097/01.sla.0000137343.63376.19. PMID 15319713
- [Background] Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007 Aug 23;357(8):741-52. doi: 10.1056/NEJMoa066254. PMID 17715408
- [Background] Cremieux PY, Buchwald H, Shikora SA, Ghosh A, Yang HE, Buessing M. A study on the economic impact of bariatric surgery. Am J Manag Care. 2008 Sep;14(9):589-96. PMID 18778174
- [Background] Santry HP, Gillen DL, Lauderdale DS. Trends in bariatric surgical procedures. JAMA. 2005 Oct 19;294(15):1909-17. doi: 10.1001/jama.294.15.1909. PMID 16234497
- [Background] Flum DR, Khan TV, Dellinger EP. Toward the rational and equitable use of bariatric surgery. JAMA. 2007 Sep 26;298(12):1442-4. doi: 10.1001/jama.298.12.1442. No abstract available. PMID 17895461
- [Background] Meguid MM, Glade MJ, Middleton FA. Weight regain after Roux-en-Y: a significant 20% complication related to PYY. Nutrition. 2008 Sep;24(9):832-42. doi: 10.1016/j.nut.2008.06.027. PMID 18725080
- [Background] Nguyen NT. Reoperations and revisions in bariatric surgery. Surg Endosc. 2007 Nov;21(11):1907-8. doi: 10.1007/s00464-007-9572-6. Epub 2007 Sep 8. No abstract available. PMID 17828427
- [Background] Sapala JA, Wood MH, Sapala MA, Flake TM Jr. Marginal ulcer after gastric bypass: a prospective 3-year study of 173 patients. Obes Surg. 1998 Oct;8(5):505-16. doi: 10.1381/096089298765554061. PMID 9819081
- [Background] Higa KD, Boone KB, Ho T. Complications of the laparoscopic Roux-en-Y gastric bypass: 1,040 patients--what have we learned? Obes Surg. 2000 Dec;10(6):509-13. doi: 10.1381/096089200321593706. PMID 11175957
- [Background] Sanyal AJ, Sugerman HJ, Kellum JM, Engle KM, Wolfe L. Stomal complications of gastric bypass: incidence and outcome of therapy. Am J Gastroenterol. 1992 Sep;87(9):1165-9. PMID 1519574
- [Background] Capella JF, Capella RF. Staple Disruption and Marginal Ulceration in Gastric Bypass Procedures for Weight Reduction. Obes Surg. 1996 Feb;6(1):44-49. doi: 10.1381/096089296765557259. PMID 10731249
- [Background] Capella JF, Capella RF. Gastro-gastric fistulas and marginal ulcers in gastric bypass procedures for weight reduction. Obes Surg. 1999 Feb;9(1):22-7; discussion 28. doi: 10.1381/096089299765553674. PMID 10065576
- [Background] Jordan JH, Hocking MP, Rout WR, Woodward ER. Marginal ulcer following gastric bypass for morbid obesity. Am Surg. 1991 May;57(5):286-8. PMID 2039124
- [Background] Sacks BC, Mattar SG, Qureshi FG, Eid GM, Collins JL, Barinas-Mitchell EJ, Schauer PR, Ramanathan RC. Incidence of marginal ulcers and the use of absorbable anastomotic sutures in laparoscopic Roux-en-Y gastric bypass. Surg Obes Relat Dis. 2006 Jan-Feb;2(1):11-6. doi: 10.1016/j.soard.2005.10.013. PMID 16925306
- [Background] Lublin M, McCoy M, Waldrep DJ. Perforating marginal ulcers after laparoscopic gastric bypass. Surg Endosc. 2006 Jan;20(1):51-4. doi: 10.1007/s00464-005-0325-0. Epub 2005 Dec 7. PMID 16333541
- [Background] St Jean MR, Dunkle-Blatter SE, Petrick AT. Laparoscopic management of perforated marginal ulcer after laparoscopic Roux-en-Y gastric bypass. Surg Obes Relat Dis. 2006 Nov-Dec;2(6):668. doi: 10.1016/j.soard.2006.09.011. No abstract available. PMID 17138240
- [Background] Chin EH, Hazzan D, Sarpel U, Herron DM. Multimedia article. Laparoscopic repair of a perforated marginal ulcer 2 years after gastric bypass. Surg Endosc. 2007 Nov;21(11):2110. doi: 10.1007/s00464-007-9486-3. Epub 2007 Aug 18. PMID 17704879
- [Background] Wheeler AA, de la Torre RA, Fearing NM. Laparoscopic repair of perforated marginal ulcer following Roux-en-Y gastric bypass: a case series. J Laparoendosc Adv Surg Tech A. 2011 Jan-Feb;21(1):57-60. doi: 10.1089/lap.2010.0402. Epub 2011 Jan 19. PMID 21247305
- [Background] Nguyen NT, Hinojosa MW, Gray J, Fayad C. Reoperation for marginal ulceration. Surg Endosc. 2007 Nov;21(11):1919-21. doi: 10.1007/s00464-007-9538-8. Epub 2007 Aug 19. No abstract available. PMID 17705072
- [Background] Patel RA, Brolin RE, Gandhi A. Revisional operations for marginal ulcer after Roux-en-Y gastric bypass. Surg Obes Relat Dis. 2009 May-Jun;5(3):317-22. doi: 10.1016/j.soard.2008.10.011. Epub 2008 Nov 6. PMID 19136312
- [Background] Hata JA, DeMaria EJ, Portenier DD, et al. Marginal ulcer after 1,792 laparoscopic Roux-en-Y gastric bypass (LRYGB) procedures: incidence, medical and surgical treatment and complications. Surg Obes Relat Dis 2008; 4:308-9 (abstract).
- [Background] Madan AK, DeArmond G, Ternovits CA, Beech DJ, Tichansky DS. Laparoscopic revision of the gastrojejunostomy for recurrent bleeding ulcers after past open revision gastric bypass. Obes Surg. 2006 Dec;16(12):1662-8. doi: 10.1381/096089206779319400. PMID 17217644
- [Background] Silver R, Levine MS, Williams NN, Rubesin SE. Using radiography to reveal chronic jejunal ischemia as a complication of gastric bypass surgery. AJR Am J Roentgenol. 2003 Nov;181(5):1365-7. doi: 10.2214/ajr.181.5.1811365. No abstract available. PMID 14573435
- [Background] Ruutiainen AT, Levine MS, Williams NN. Giant jejunal ulcers after Roux-en-Y gastric bypass. Abdom Imaging. 2008 Sep-Oct;33(5):575-8. doi: 10.1007/s00261-007-9344-8. PMID 18175166
- [Background] Wallace JL. Pathogenesis of NSAID-induced gastroduodenal mucosal injury. Best Pract Res Clin Gastroenterol. 2001 Oct;15(5):691-703. doi: 10.1053/bega.2001.0229. PMID 11566035
- [Background] Ben-Meir A, Sonpal I, Patterson L, et al. Cigarette smoking, but not NSAID or alcohol use of comorbidities, is associated with anastomotic ulcer in Roux-en-Y gastric bypass (RYGB) patients. Surg Obes Relat Dis 2005;1: 263-4.
- [Background] Kurata JH, Nogawa AN. Meta-analysis of risk factors for peptic ulcer. Nonsteroidal antiinflammatory drugs, Helicobacter pylori, and smoking. J Clin Gastroenterol. 1997 Jan;24(1):2-17. doi: 10.1097/00004836-199701000-00002. PMID 9013343
- [Background] Schreiber H, Ben-Meir A, Sonpal I, et al. Cigarette smoking, but not the presence of H.pylori, is associated with anastomotic ulcers in Roux-en-Y gastric bypass patients. Surg Obes Relat Dis 2005;1:257.
- [Background] Huang JQ, Sridhar S, Hunt RH. Role of Helicobacter pylori infection and non-steroidal anti-inflammatory drugs in peptic-ulcer disease: a meta-analysis. Lancet. 2002 Jan 5;359(9300):14-22. doi: 10.1016/S0140-6736(02)07273-2. PMID 11809181
- [Background] Yang CS, Lee WJ, Wang HH, Huang SP, Lin JT, Wu MS. The influence of Helicobacter pylori infection on the development of gastric ulcer in symptomatic patients after bariatric surgery. Obes Surg. 2006 Jun;16(6):735-9. doi: 10.1381/096089206777346754. PMID 16756734
- [Background] Papasavas PK, Gagne DJ, Donnelly PE, Salgado J, Urbandt JE, Burton KK, Caushaj PF. Prevalence of Helicobacter pylori infection and value of preoperative testing and treatment in patients undergoing laparoscopic Roux-en-Y gastric bypass. Surg Obes Relat Dis. 2008 May-Jun;4(3):383-8. doi: 10.1016/j.soard.2007.08.014. Epub 2007 Nov 5. PMID 17974495
- [Background] Teyssen S, Singer MV. Alcohol-related diseases of the oesophagus and stomach. Best Pract Res Clin Gastroenterol. 2003 Aug;17(4):557-73. doi: 10.1016/s1521-6918(03)00049-0. PMID 12828955
- [Background] Bode C, Bode JC. Effect of alcohol consumption on the gut. Best Pract Res Clin Gastroenterol. 2003 Aug;17(4):575-92. doi: 10.1016/s1521-6918(03)00034-9. PMID 12828956
- [Background] Glauser J, Queen JR. An overview of non-cardiac cocaine toxicity. J Emerg Med. 2007 Feb;32(2):181-6. doi: 10.1016/j.jemermed.2006.05.044. Epub 2007 Jan 22. PMID 17307630
- [Background] Lee HS, LaMaute HR, Pizzi WF, Picard DL, Luks FI. Acute gastroduodenal perforations associated with use of crack. Ann Surg. 1990 Jan;211(1):15-7. doi: 10.1097/00000658-199001000-00003. PMID 2403771
- [Background] Arrillaga A, Sosa JL, Najjar R. Laparoscopic patching of crack cocaine-induced perforated ulcers. Am Surg. 1996 Dec;62(12):1007-9. PMID 8955237
- [Background] Sharma R, Organ CH Jr, Hirvela ER, Henderson VJ. Clinical observation of the temporal association between crack cocaine and duodenal ulcer perforation. Am J Surg. 1997 Dec;174(6):629-32; discussion 632-3. doi: 10.1016/s0002-9610(97)00215-8. PMID 9409587
- [Background] Schuster KM, Feuer WJ, Barquist ES. Outcomes of cocaine-induced gastric perforations repaired with an omental patch. J Gastrointest Surg. 2007 Nov;11(11):1560-3. doi: 10.1007/s11605-007-0257-1. Epub 2007 Aug 15. PMID 17701263
- [Background] Mason EE. Warning patients about cocaine and aspirin. Obes Surg. 1998 Jun;8(3):312-3. doi: 10.1381/096089298765554539. No abstract available. PMID 9678199
- [Background] Steinberg KP. Stress-related mucosal disease in the critically ill patient: risk factors and strategies to prevent stress-related bleeding in the intensive care unit. Crit Care Med. 2002 Jun;30(6 Suppl):S362-4. doi: 10.1097/00003246-200206001-00005. PMID 12072662
- [Background] Spirt MJ. Stress-related mucosal disease: risk factors and prophylactic therapy. Clin Ther. 2004 Feb;26(2):197-213. doi: 10.1016/s0149-2918(04)90019-7. PMID 15038943
- See also: "Click here for more information about the department sponsor´s web site" — http://www.fresno.ucsf.edu/surgery/